CLINICAL TRIAL: NCT03449992
Title: The Effects of Beet-root Juice Supplementation on Exercise Economy, Rating of Perceived Exertion and Running Mechanics in Elite Distance Runners
Brief Title: The Effects of Nitrate Supplementation on Elite Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Camilo Jose Cela University (Other); Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Carlos Balsalobre-Fernández, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BEETRUN
Record Dates: First submitted 2018-02-19; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Nutrition; Physical Performance; Sport Physiology; Nitrates; Elite Athletes

STUDY DESIGN:
Intervention Model Description: Twelve elite distance runners were randomly assigned to either an intervention group or a placebo group. Participants in each group consumed beetroot juice or a placebo drink for 15 consecutive days.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Twelve participants were randomly assigned to either an intervention group or a placebo group, and a 4 digits code based on their Spanish ID card were used to code their names.
  Then, an independent researcher prepared individual bags with either a 15-days worth of placebo drinks or beetroot drinks, and gave it to the athletes. Then, this person was withdrawn for the research procedures.
  Finally, another group of researchers, without knowing what athlete was on each group (intervention or placebo), conducted the performance tests pre and post 15 days of supplementation, and another group analyzed the data once collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this group ingested nitrate-rich beetroot juice for 15 days
  Interventions: Dietary Supplement: nitrate-rich beetroot juice
- Placebo group (Placebo Comparator): Participants in this group ingested a placebo drink for 15 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: nitrate-rich beetroot juice — Nitrate-rich beetroot juice supplementation was administered for 15 consecutive days to participants in this arm
  Other Names: Beetroot juice
  Arms: Intervention group
Dietary Supplement: Placebo — Placebo drink
  Arms: Placebo group

SUMMARY:
This study analyzed the effects of 15 days of beetroot juice supplementation on different performance measures in elite Spanish distance runners

DETAILED DESCRIPTION:
This study analyzed the effects of 15 days beetroot juice supplementation on the VO2max, running economy, exercise perceived exertion, muscle power and locomotion mechanics in a group of 12 elite Spanish middle and long distance runners

ELIGIBILITY:
Inclusion Criteria:

* Competing in national and international events
* Personal best in urban 10k: 33 minutes 0 seconds

Exclusion Criteria:

* Injury

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Running economy | Changes from baseline at 15 days
  The cost of running (oxygen consumption) at different speeds

SECONDARY OUTCOMES:
Time to exhaustion | Changes from baseline at 15 days
  Time that the athlete endured running until voluntarily ending the exercise
Muscle power | Changes from baseline at 15 days
  Ability to produce muscle power in a jump test
Muscle oxygenation | Changes from baseline at 15 days
  Saturation of O2 in the vastus lateralis during exercise
RPE | Changes from baseline at 15 days
  Rate of perceived exertion during the exercise
Running mechanics | Changes from baseline at 15 days
  Contact and flight time of each step during the exercise

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Balsalobre-Fernández, PhD, Principal Investigator — Universidad Autonoma de Madrid

IPD SHARING:
Plan to Share IPD: Yes
Coded database with data of the pre-post measures will be made available
Supporting Information: Analytic Code
Time Frame: Indefinitely available
Access Criteria: Open access
URL: https://doi.org/10.6084/m9.figshare.5873190.v1

REFERENCES:
- Available data/document: Individual Participant Data Set — https://doi.org/10.6084/m9.figshare.5873190.v1